CLINICAL TRIAL: NCT03176862
Title: Onset and Functional Consequences of Left Ventricular (LV) Fibrosis in Chronic Kidney
Brief Title: Left Ventricular Fibrosis in Chronic Kidney Disease
Acronym: FibroCKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Manvir Kaur Hayer (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Dr Manvir Kaur Hayer, Clinical Research Fellow, University Hospital Birmingham NHS Foundation Trust
Organization: University Hospital Birmingham NHS Foundation Trust (Other)
Other Study IDs: UHB
Record Dates: First submitted 2017-05-18; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Diseases; Cardio-Renal Syndrome; Myocardial Fibrosis; Uraemic Cardiomyopathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardio-Renal Syndrome | interventions — Exercise Test; Echocardiography, Stress; Electrocardiography; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CKD: 40 patients per group of CKD from stage 2 to stage 5.
  Interventions: Diagnostic Test: cardiac magnetic resonance scan; Diagnostic Test: Cardiopulmonary exercise test with stress echocardiogram; Diagnostic Test: 24-hour ECG holter monitor; Diagnostic Test: 12-lead ECG; Biological: Blood test
- Kidney transplant recipients: 20 live-donor recipients will be studied pre-operatively and then followed up at 6 weeks and 1 years post-operatively.
  Interventions: Diagnostic Test: cardiac magnetic resonance scan; Diagnostic Test: 24-hour ECG holter monitor; Diagnostic Test: 12-lead ECG; Diagnostic Test: Cardiopulmonary exercise test; Biological: Blood test
- Controls: 40 healthy controls and 40 hypertensive controls.
  Interventions: Diagnostic Test: cardiac magnetic resonance scan; Diagnostic Test: Cardiopulmonary exercise test with stress echocardiogram; Diagnostic Test: 12-lead ECG; Diagnostic Test: Cardiopulmonary exercise test; Biological: Blood test

INTERVENTIONS:
Diagnostic Test: cardiac magnetic resonance scan — An MRI scan of the heart
Diagnostic Test: Cardiopulmonary exercise test with stress echocardiogram — An exercise bicycle test with echocardiogram done during the exercise.
  Groups: CKD; Controls
Diagnostic Test: 24-hour ECG holter monitor — 3 stickers attached to a small monitor are worn for 24 hours.
  Groups: CKD; Kidney transplant recipients
Diagnostic Test: 12-lead ECG — Can be done immediately by the bedside.
Diagnostic Test: Cardiopulmonary exercise test — An exercise bicycle test. No stress echocardiogram.
  Groups: Controls; Kidney transplant recipients
Biological: Blood test — 20 mls of blood will be taken to measure routine laboratory tests and biomarkers of fibrosis.

SUMMARY:
This study aims to understand the onset an functional consequences of left ventricular interstitial fibrosis in patients with chronic kidney disease (stage 2 to 5), as well as assess whether transplantation results in a regression of cardiac fibrosis.Thus all patients will undergo: 1) a cardiac magnetic resonance imaging (MRI) scan to assess cardiac function and measure left ventricular interstitial fibrosis; 2) a cardiopulmonary stress echocardiogram to understand the functional consequences of fibrosis and rule out any underlying ischaemic heart disease; 3) a 24 hour holter monitor and electrocardiogram (ECG) to assess whether these patients are at higher risk of arrhythmia.

DETAILED DESCRIPTION:
Aim and objectives:

The primary objective of this study is to test the following hypotheses:

i) Patients with early stage chronic kidney disease (CKD) exhibit diffuse LV fibrosis manifest by prolonged native myocardial T1 times and expansion of the extracellular volume (ECV) measured on MRI with a graded relationship to eGFR (stage of CKD), independent of blood pressure and arterial stiffness.

The secondary research objectives are to test the following hypotheses:

i) Prolonged native myocardial T1 times are associated with impaired diastolic function, altered arterial-ventricular interaction and impaired effort tolerance.

ii) Prolonged T1 times correlate with increases in serum biomarkers of collagen turnover associated with myocardial fibrosis that could be used to risk stratify individuals and enable targeted, personalized clinical care.

iii) Renal transplantation results in a regression of myocardial fibrosis as measured by T1 mapping.

DESIGN:

A cross-sectional analysis of 40 patients in each stage 2-5 CKD will be undertaken. These individuals will only be studied once (at baseline). In addition to this, at least 20 patients will be studied who are about to undergo a kidney transplant. These individuals will be studied at baseline (around the time of surgery), at 6 weeks post-operatively, and then 1 year post-operatively to assess the effect on renal transplantation on myocardial fibrosis.

SUBJECTS:

Patients will be recruited from the clinics run by University Hospitals Birmingham NHS Foundation Trust (UHB) with stages 2, 3, 4 and 5 CKD defined using eGFR calculated with the 4-variable 'Modification of Diet in Renal Disease' (MDRD) equation, with a minimum of two consecutive tests at least 90 days apart. Forty patients will be recruited per group of CKD. All study subjects will undergo a cardiac MRI scan, a cardiopulmonary exercise tests with stress echocardiogram, a 24-hour ECG holter monitor, and blood tests.

CONTROLS:

Forty healthy control subjects and forty hypertensive control subjects will be studied. All patients will undergo the identical research protocol to the CKD subjects, except they will not have a stress echocardiogram or an ECG holter monitor.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* CKD stage 2, 3, 4 and 5

Exclusion Criteria:

* Pregnancy
* Ischaemic heart disease (angina, ACS)
* Cerebral vascular disease
* Peripheral vascular disease
* Renovascular disease
* Diabetes mellitus
* Valvular heart disease (more than mild)
* Established diagnosis of heart failure
* Cannot have an MRI scan

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable CKD from early to severe late stage (stage 2 to 5). Patients expected to undergo live-donor kidney transplantation. Healthy controls. Hypertensive controls (stable, well controlled hypertension).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The effect of eGFR on heart muscle scarring (measured from cardiac MRI using T1 times). | One baseline visit only
  eGFR is a measurement of kidney function. Heart muscle scarring levels can be derived from cardiac MRI using a technique called T1 mapping. T1 maps of the heart will be acquired using cardiac MRI. eGFR will be measured from a blood tests, using the MDRD equation. The relationship between the measured T1 times and eGFR will be analysed using statistical tests.

SECONDARY OUTCOMES:
The relationship between prolonged myocardial T1 and diastolic function. | One baseline visit only
  The following diastolic function parameters will be measured on echocardiography: E/A, deceleration time and E/e'.
The relationship between prolonged myocardial T1 and effort tolerance. | One baseline visit only
  The percent predicted peak oxygen uptake during exercise testing will be used as a surrogate marker of effort tolerance.
The effect of renal transplantation on myocardial fibrosis. | Baseline visit (pre-operation), then follow up at 6 weeks and 1 year.
  Myocardial T1 times (cardiac MRI) and eGFR (blood testing) will best measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola C Edwards, PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hayer MK, Radhakrishnan A, Price AM, Liu B, Baig S, Weston CJ, Biasiolli L, Ferro CJ, Townend JN, Steeds RP, Edwards NC; Birmingham Cardio-Renal Group. Defining Myocardial Abnormalities Across the Stages of Chronic Kidney Disease: A Cardiac Magnetic Resonance Imaging Study. JACC Cardiovasc Imaging. 2020 Nov;13(11):2357-2367. doi: 10.1016/j.jcmg.2020.04.021. Epub 2020 Jul 15. PMID 32682713